CLINICAL TRIAL: NCT03108573
Title: Improved Detection of Multiple Sclerosis Plaques in Inversion Recovery by Optimization of Sequence Parameters
Acronym: FLAIR-SEP
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SC/DM_JSY_2012-3
Record Dates: First submitted 2017-03-16; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates different optimized MRI sequences for the detection of brain lesions in patients with multiple sclerosis in comparison with the recommended FLAIR sequence

DETAILED DESCRIPTION:
MRI is a tool of choice for detecting demyelinating lesions in Multiple Sclerosis (MS) disease. On a consensual basis, the detection of those lesions in done on FLAIR (FLuid Attenuated Inversion Recovery) sequences, weighted T2 with cancelling of fluid signal, leading to a much better contrast between the lesion and the environment. The environment is displayed as a iso-signal for the surrounding healthy brain's white matter and as a hypo-signal for the fluids. Keys parameters indicative of the sequence's contrast are the echo time, the reversal time, and the repetition time, wich seems to be crucial to detect the lesions, according to relatively discordant results of publications using different technologies of FLAIR. Although 3D FLAIR sequences play an essential role for diagnosis and evaluation (evolution under treatment, prognosis) of demyelinating pathologies there is no consensus on parameters used on routine basis.

The aim of the trial is to discover the optimal combination of theses parameters so as to well detect the lesions.

ELIGIBILITY:
Inclusion Criteria:

* relapsing remitting multiple sclerosis
* MRI required

Exclusion Criteria:

* MRI contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a definite diagnosis of multiple sclerosis, with a follow-up MRI
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
Number of detectable lesions | baseline
  quantification of lesions on each sequence

SECONDARY OUTCOMES:
localisation of lesions | baseline
  proportion of lesions localised in cerebellum or brainstem, on each sequence